CLINICAL TRIAL: NCT06899685
Title: KINESIOTAPING VERSUS INSTRUMENT ASSISTED SOFT TISSUE MOBILIZATION ON UPPER TRAPEZIUS MYOFASCIAL TRIGGER POINTS: A RANDOMIZED CONTROLLED TRIAL Kinesiotaping (KT) is a Non-invasive Method to Treat Musculoskeletal Disorders. it is Non-invasive, Painless, and Less Time-consuming Than Other Options With Fewer Side Effects. IASTM is a Traditional Chinese Therapy Known as "Guasha". IASTM is a Simple and Practical Technique
Brief Title: KT vs IASTM on Upper Trapezius Myofascial Trigger Points To Compare Effect of KT VS IASTM on Pain Intensity, Pain Pressure Threshold, Cervical Range of Motion and Functional Disability Level.
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Reham Sayed Mesaed (Other)
Responsible Party: Sponsor-Investigator, Reham Sayed Mesaed, Master's Student Researcher, Cairo University
Organization: Cairo University (Other)
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: P.T.REC/012/004971
Record Dates: First submitted 2025-03-21; First posted 2025-03-28 (Actual); Last update posted 2025-03-28 (Actual); Status verified 2024-06

CONDITIONS: Myofacial Pain Syndromes
MeSH Terms: conditions — Facial Neuralgia

STUDY DESIGN:
Who Masked: Participant, Care Provider
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: Yes

ARMS (3):
- tradional physical therapy (Active Comparator): This group received traditional therapy( Instructions, hot backs, Deep transverse friction massage, passive &self stretch, Neck isometric and Scapular retraction exercises) (three sessions per week for 4 weeks).
  Interventions: Other: tradional physical therapy treatment
- Kinesiotaping (Experimental): This group received KT in addition to Traditional physical therapy program (two sessions per week for 4 weeks).
  Interventions: Other: tradional physical therapy treatment; Other: KT
- IASTM (Experimental): This group received IASTM in addition to Traditional physical therapy program (three sessions per week for 4 weeks).
  Interventions: Other: tradional physical therapy treatment; Device: IASTM

INTERVENTIONS:
Other: tradional physical therapy treatment — Instructions, hot backs, Deep transverse friction massage, passive &self stretch, Neck isometric and Scapular retraction exercises
Other: KT — Kinesiotaping
  Arms: Kinesiotaping
Device: IASTM — Instrument Assisted Soft Tissue Mobolization
  Arms: IASTM

SUMMARY:
This study would answer the following question: Is there a difference in the effects between IASTM and KT on pain intensity level, pain pressure threshold, cervical range of motion (ROM), functional disability level and satisfaction level in subjects with upper trapezius myofascial trigger points?

The aims of this study are:

1. To investigate the effect of KT and IASTM on pain intensity level in subjects with upper trapezius myofascial trigger points.
2. To investigate the effects of KT and IASTM on pain pressure threshold in subjects with upper trapezius myofascial trigger points.
3. To investigate the effects of KT and IASTM on cervical range of motion (ROM) in subjects with myofascial trigger points.
4. To investigate the effect of KT and IASTM on functional disability level in subjects with upper trapezius myofascial trigger points.
5. To investigate the effects of KT and IASTM on satisfaction level in subjects with myofascial trigger points.

ELIGIBILITY:
Inclusion Criteria:

- 1) Fifty subjects with age ranged from 18 to 23 years old (Formen et al., 2014).

2) From both genders with normal BMI ranges between 18.5:24.9 kg/m2. Had MTrPs of unilateral UT muscle (Shamseldeen et al., 2023).

Exclusion Criteria:

* 1. History of whiplash injury (Emshi et al., 2021). 2. History of head, neck, cervical spine or shoulder surgery (Emshi., et al 2021) 3. History of cervical radiculopathy (Emshi et al., 2021) 4. Patients with malignancy (Shamseldeen et al., 2023). 5. Cervical spine fractures (Shamseldeen et al., 2023). 6. Myelopathy (Shamseldeen et al., 2023). 7. Having undergone physical therapy within the past three months before the study.

  8. Non - rheumatologic diseases as multiple sclerosis, thyroid dysfunction and chronic infection.

  9. Rheumatologic condition as poly-articular osteoarthritis, rheumatoid arthritis and advanced cervical spine degenerative diseases.

  10. Presence of skin diseases (Luz Júnior et al., 2015). 11. Pregnancy (Luz Júnior et al., 2015).

Ages: 19 Years to 23 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 50 (Estimated)
Dates: Start 2024-08-01 (Actual); Primary Completion 2024-09-01 (Actual); Study Completion 2025-04-01 (Estimated)

PRIMARY OUTCOMES:
KT vs IASTM on upper trapezius myofascial trigger points | one month
pain intensity level | change at pain intensity level through 4 weeks
  pain intensity level of neck pain

SECONDARY OUTCOMES:
pain pressure threshold | change at pain pressure threshold through 4 weeks
  pain pressure threshold of neck pain
cervical range of motion | change at cervical range of motion through 4 weeks
  range of motion of cervical spine

OTHER OUTCOMES:
functional disability level | change at functional disability level through 4 weeks
  functional disability level by Arabic Neck Disability Index

CONTACTS AND LOCATIONS:
Locations (1):
- Clinic, Banī Suwayf, Egypt